CLINICAL TRIAL: NCT01123265
Title: Dendritic Cell-Specific Transmembrane Protein (DC-STAMP) as a Severity and Response Biomarker in Psoriatic Arthritis
Brief Title: National Psoriasis Foundation - Dendritic Cell-Specific Transmembrane Protein (DC-Stamp) Biomarker Study
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Psoriasis Foundation (Other)
Responsible Party: Principal Investigator, Christopher Ritchlin, M.D., M.P.H.; Professor of Medicine Allergy, Immunology & Rheumatology Division, University of Rochester
Other Study IDs: RSRB - 32368
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Psoriatic Arthritis
Keywords: PsA; methotrexate; Anti-TNF; TNF; DC-Stamp
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anti-TNF
  Interventions: Drug: Anti-TNF
- Methotrexate
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Subjects will start Methotrexate which will be escalated from 7.5 mg weekly to 15 mg/weekly over a 3 week period.
  Groups: Methotrexate
Drug: Anti-TNF — Anti-TNF to be administered per standard of care within the practice.
  Groups: Anti-TNF

SUMMARY:
The purpose of this study is to determine whether DC-STAMP, a protein on the surface of osteoclast precursors (OCPs), can be used as a biologic marker in Psoriatic Arthritis (PsA). With this marker the investigators hope to learn more about how OCPs develop as well as find out if DC-STAMP predicts PsA severity and how well treatment works in PsA.

DETAILED DESCRIPTION:
Psoriatic Arthritis (PsA), a phenotypically heterogeneous disorder, is characterized by joint damage observed in over half of the patients with early disease. While anti-tumor necrosis factor (TNF) agents have greatly improved signs and symptoms and lessened joint damage, the fact that only a fraction of patients achieve complete remission underscores the tremendous unmet need for this population. To date, a biomarker that can stratify patients by severity and can serve as a leading indicator of treatment response has not been identified.

Our laboratory demonstrated that circulating osteoclast precursors (OCP) are elevated in PsA patients. OCP decline rapidly following anti-TNF therapy and levels are higher in subjects with erosive arthritis compared to those with no x-ray changes. The OCP are derived from CD14+ monocytes and the assay entails culture techniques that are costly, expensive and labor intensive. We developed an antibody (1A2) to Dendritic Cell Specific Transmembrane Protein (DC-STAMP), a potential marker of the OCP population, for analysis by flow cytometry. We found that: 1) the level of monocyte DC-STAMP expression correlated with in vitro osteoclast formation; 2) DC-STAMP expression is significantly elevated in PBMC from PsA subjects compared to controls; 3) TNF dramatically upregulated the expression of DC-STAMP in vitro; 4) DC-STAMP surface expression declined following anti-TNF therapy; 5) subsets of CD3+ cells also express DC-STAMP on the cell membrane. Based on these preliminary data, three hypotheses are proposed:

1. DC-STAMP+ CD3+ T cells belong to the Th17 subset which facilitates OC generation;
2. DC-STAMP is a marker of disease severity in PsA;
3. DC-STAMP is a biomarker of treatment response in PsA.

We propose three Specific Aims to test these hypotheses.

Aim 1 To examine whether DC-STAMP+CD3+ cells belong to the Th17 cell subset, PBMC will be stained with Th17-specific antibodies in PsA subjects with elevated DC-STAMP expression. We will also examine the role of T cells in osteoclastogenesis directly by co-culture experiments and we will use monocyte cultures without added lymphocytes as controls. The expression of DC-STAMP on circulating dendritic cells will be examined ex vivo with 11-color flow cytometry.

Aim 2 To determine if increased DC-STAMP expression is associated with more severe features of PsA, DC-STAMP expression in 40 PsA subjects will be determined and correlated with clinical variables of arthritis and skin disease, CRP and x-ray damage.

Aim 3 To examine if DC-STAMP is a response marker to anti-TNF treatment, we will recruit 20 PsA patients in Aim 2 with elevated DC-STAMP expression and divide them into 2 groups. Ten subjects will receive methotrexate, and ten will receive anti-TNF therapy. The correlation between DC-STAMP variables (percentage of 1A2+ divided by 1A2 - cells X 100) and the variables detailed in Aim 2 will be analyzed in these 2 treatment groups at 2 different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be >18 years old
2. Subject must have >3 tender and swollen joints
3. Subject must have must have a target lesion of greater than 3 cm in diameter
4. Subjects who meet the the ClASsification of Psoriatic ARthritis (CASPAR) criteria for PsA
5. Subjects must have a DC-STAMP pattern III or IV

Exclusion Criteria:

1. Subjects with active inflammatory synovitis, dactylitis, enthesitis, osteoarthritis, axial disease, Subjects with a SLE, Sjogren's syndrome, scleroderma or inflammatory muscle disease
2. Subjects with an active malignancy
3. Subjects currently on biologic agents (anti-TNF agents, anti-T or B cells agents) and/or disease-modifying antirheumatic drugs (DMARDs) (methotrexate, leflunomide, hydroxychloroquine, azulfidine, cyclosporine, azathioprine)
4. Subjects who have been off DMARDs or biologics for less than 3 months
5. Subjects judged ineligible at the discretion of the PI
6. Subjects with a history of crystalline arthritis (gout, pseudogout)
7. Subject pregnancy or breast feeding
8. History of recurrent infections - AIM 3 Specific
9. Demyelinating disorders - AIM 3 Specific
10. Prior non-responsiveness to TNFi - AIM 3 Specific
11. Subjects who have a BMI >30 - AIM 3 Specific MTX arm
12. Subjects who have a history of type II diabetes - AIM 3 Specific MTX arm
13. Subjects with a history of substance abuse including alcohol - AIM 3 Specific MTX arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female population that are 18 years old and older.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Analysis of T cell subset and dendritic cell (DC) subset for DC-STAMP expression | Week 0 (Baseline)
  Determine whether DC-STAMP+ cells belong to the Th17 subset and also analyze the DC subsets for DC-STAMP expression.
Analysis of T cell subset and DC subset for DC-STAMP expression | Week 16
  Determine whether DC-STAMP+ cells belong to the Th17 subset and also analyze the DC subsets for DC-STAMP expression.
DC-STAMP as a marker of disease severity in PsA | Week 0 (Baseline)
  Baseline measurement of DC-STAMP expression will be collected in order to assist in determining whether it is associated with more severe features of PsA. DC-STAMP expression will be correlated with clinical variables of arthritis and skin disease, CRP and x-ray damage.
DC-STAMP as a marker of disease severity in PsA | Week 16
  Measurement of DC-STAMP expression will be collected in order to assist in determining whether it is associated with more severe features of PsA. DC-STAMP expression will be correlated with clinical variables of arthritis and skin disease, CRP and x-ray damage.
DC-STAMP as a biomarker of treatment response in PsA | Week 0 (Baseline)
  A baseline measurement of DC-STAMP as a response marker to treatment will be collected. Ten subjects will receive methotrexate and ten will receive anti-TNF therapy. The correlation between DC-STAMP variables (percentage of 1A2+ divided by 1A2 - cells X 100) and the variables detailed in Aim 2 will be analyzed in these 2 treatment groups at 2 different time points.
DC-STAMP as a biomarker of treatment response in PsA | Week 16
  A measurement of DC-STAMP as a response marker to treatment will be collected. Ten subjects received methotrexate and ten received anti-TNF therapy. The correlation between DC-STAMP variables (percentage of 1A2+ divided by 1A2 - cells X 100) and the variables detailed in Aim 2 will be analyzed in these 2 treatment groups at 2 different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD / MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States